CLINICAL TRIAL: NCT02168972
Title: A Prospective, Non-randomized Clinical Study to Assess Safety and Performance of a Device for Global Mapping and Ablation of the Left Atrium for the Treatment of Atrial Fibrillation
Brief Title: Safety and Performance of a GLOBAL Mapping and Ablation Device for the Treatment of Atrial Fibrillation (GLOBAL-AF)
Acronym: GLOBAL-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kardium Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOC-19996
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; global; radiofrequency RF ablation; left atrium anatomical and electrophysiological mapping
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Global mapping and ablation device (Experimental)
  Interventions: Device: Global mapping and ablation device

INTERVENTIONS:
Device: Global mapping and ablation device — During the procedure the Globe catheter will be delivered via standard femoral vein access and transseptal puncture. Anatomical and electrophysiological mapping of the LA will be followed by pulmonary vein isolation (PVI) by RF ablation. Additional lesions will be created as deemed appropriate by the investigator.
  Other Names: Globe® Mapping and Ablation System

SUMMARY:
The purpose of this study is to provide clinical data pertaining to the safety and performance of the Globe® Mapping and Ablation System for treating patients with atrial fibrillation.

DETAILED DESCRIPTION:
Upon successful enrolment, subjects will be scheduled for mapping and radiofrequency (RF) ablation. Cardiac CT imaging, echocardiography and baseline 12-lead ECG will be performed pre-procedure for screening and health assessment. During the procedure the Globe catheter will be delivered via standard femoral vein access and transseptal puncture. Anatomical and electrophysiological mapping of the left atrium (LA) will be followed by RF ablation to achieve pulmonary vein isolation (PVI). Additional lesions will be created as deemed appropriate by the investigator. Intracardiac electrogram mapping will be used to confirm PVI during the procedure. Echocardiography will be performed at discharge to assess cardiac function. Electrocardiograms by 12-lead ECG and 7-day Holter monitoring will be recorded at discharge, and 3, 6 and 12 months after treatment. Follow-up assessments will be performed at discharge, 7 days, and 1, 3, 6 and 12 months after treatment, to track freedom from documented AF and adverse events. Subject-reported AF symptomology and quality of life will also be assessed during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for ablation, with a documented history of symptomatic paroxysmal atrial fibrillation
* Between 18 and 80 years of age, inclusive

Exclusion Criteria:

* Patients who have contraindications to open heart surgery
* Patients from an Intensive Care Unit
* Patients requiring concurrent right atrial ablation or who have had previous left atrial ablation
* Previous cardiac procedure or known abnormalities that would interfere with device delivery, position, or treatment efficacy
* History of a documented thromboembolic event or bleeding abnormalities
* Contraindication to anticoagulation therapy
* Mental impairment or other conditions, which may not allow patient to understand the nature, significance and scope of the study
* Anatomy that would prevent safe and appropriate introduction or delivery of the Globe device into the patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Rate of subjects presenting pre-defined serious adverse events occurring within 7 days of the procedure | 7 days
  Rate of subjects presenting with one or more of the following serious adverse events occurring within 7-days of the procedure:
  * Transient ischemic attack
  * Cerebrovascular accident
  * Major bleeding
  * Cardiac tamponade
  * Pulmonary vein stenosis
  * Pericarditis
  * Myocardial infarction
  * Diaphragmatic paralysis
  * Atrio-esophageal fistula
  * Valvular damage
  * Phrenic nerve palsy
  * Intra-procedural device complication requiring open chest or heart surgery
  * Death

SECONDARY OUTCOMES:
Subjects presenting with adverse events | Up to 1 year
  * Subjects presenting with primary serious adverse events up to 1 year
  * Subjects presenting with adverse events or serious adverse events up to 1 year
Acute procedural success | Intra-procedurally
  Acute device performance in achieving entrance block of the pulmonary veins
Rate of freedom from documented atrial fibrillation | Between 3 months and 1 year
  Rate of freedom from electrocardiographically documented atrial fibrillation between 3 months and 1 year post-ablation
Change in Quality of life and AF symptom frequency and severity scores | Up to 1 year
  Change of quality of life (SF-36) and AF symptom frequency and severity (Bubien et al 1993) questionnaire scores from baseline to 1 year after ablation

OTHER OUTCOMES:
Procedure time | Intra-procedurally
  Procedure time
Repeat ablation rate | Up to 1 year
  Rate of repeat ablation with a third party catheter or the Globe system
Fluoroscopy time and dose area product | Intra-procedurally
  Fluoroscopy time and dose area product during the procedure
Device functionality | Intra-procedurally
  Rate of procedures terminated or switched to a third-party ablation catheter due to Globe device failures

CONTACTS AND LOCATIONS:
Overall Officials: Hans Kottkamp, Prof.Dr.med., Principal Investigator — Klinik Hirslanden, Zurich
Locations (2):
- Herzzentrum Leipzig GmbH, Leipzig, Saxony, Germany
- Klinik Hirslanden, Zurich, Switzerland

REFERENCES:
- [Background] Calkins H, Kuck KH, Cappato R, Brugada J, Camm AJ, Chen SA, Crijns HJ, Damiano RJ Jr, Davies DW, DiMarco J, Edgerton J, Ellenbogen K, Ezekowitz MD, Haines DE, Haissaguerre M, Hindricks G, Iesaka Y, Jackman W, Jalife J, Jais P, Kalman J, Keane D, Kim YH, Kirchhof P, Klein G, Kottkamp H, Kumagai K, Lindsay BD, Mansour M, Marchlinski FE, McCarthy PM, Mont JL, Morady F, Nademanee K, Nakagawa H, Natale A, Nattel S, Packer DL, Pappone C, Prystowsky E, Raviele A, Reddy V, Ruskin JN, Shemin RJ, Tsao HM, Wilber D; Heart Rhythm Society Task Force on Catheter and Surgical Ablation of Atrial Fibrillation. 2012 HRS/EHRA/ECAS expert consensus statement on catheter and surgical ablation of atrial fibrillation: recommendations for patient selection, procedural techniques, patient management and follow-up, definitions, endpoints, and research trial design: a report of the Heart Rhythm Society (HRS) Task Force on Catheter and Surgical Ablation of Atrial Fibrillation. Developed in partnership with the European Heart Rhythm Association (EHRA), a registered branch of the European Society of Cardiology (ESC) and the European Cardiac Arrhythmia Society (ECAS); and in collaboration with the American College of Cardiology (ACC), American Heart Association (AHA), the Asia Pacific Heart Rhythm Society (APHRS), and the Society of Thoracic Surgeons (STS). Endorsed by the governing bodies of the American College of Cardiology Foundation, the American Heart Association, the European Cardiac Arrhythmia Society, the European Heart Rhythm Association, the Society of Thoracic Surgeons, the Asia Pacific Heart Rhythm Society, and the Heart Rhythm Society. Heart Rhythm. 2012 Apr;9(4):632-696.e21. doi: 10.1016/j.hrthm.2011.12.016. Epub 2012 Mar 1. No abstract available. PMID 22386883
- [Background] Cappato R, Calkins H, Chen SA, Davies W, Iesaka Y, Kalman J, Kim YH, Klein G, Natale A, Packer D, Skanes A, Ambrogi F, Biganzoli E. Updated worldwide survey on the methods, efficacy, and safety of catheter ablation for human atrial fibrillation. Circ Arrhythm Electrophysiol. 2010 Feb;3(1):32-8. doi: 10.1161/CIRCEP.109.859116. Epub 2009 Dec 7. PMID 19995881
- [Background] European Heart Rhythm Association; Heart Rhythm Society; Fuster V, Ryden LE, Cannom DS, Crijns HJ, Curtis AB, Ellenbogen KA, Halperin JL, Le Heuzey JY, Kay GN, Lowe JE, Olsson SB, Prystowsky EN, Tamargo JL, Wann S, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Hunt SA, Nishimura R, Ornato JP, Page RL, Riegel B, Priori SG, Blanc JJ, Budaj A, Camm AJ, Dean V, Deckers JW, Despres C, Dickstein K, Lekakis J, McGregor K, Metra M, Morais J, Osterspey A, Zamorano JL; American College of Cardiology; American Heart Association Task Force on Practice Guidelines; European Society of Cardiology Committee for Practice Guidelines; Writing Committee to Revise the 2001 Guidelines for the Management of Patients With Atrial Fibrillation. ACC/AHA/ESC 2006 guidelines for the management of patients with atrial fibrillation--executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the European Society of Cardiology Committee for Practice Guidelines (Writing Committee to Revise the 2001 Guidelines for the Management of Patients With Atrial Fibrillation). J Am Coll Cardiol. 2006 Aug 15;48(4):854-906. doi: 10.1016/j.jacc.2006.07.009. No abstract available. PMID 16904574